CLINICAL TRIAL: NCT04640896
Title: Comparison of Trigger Point Injections Versus Traditional Therapies in the Management of Postsurgical Pain in Patients Who Had Anterior Cervical Surgery
Brief Title: Trigger Point Injections in Anterior Cervical Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Anita Vincent, Assistant Professor of Anesthesiology and Critical Care, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCR191932
Record Dates: First submitted 2020-11-13; First posted 2020-11-23 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Myofacial Pain; Pain, Neck; Pain, Back; Cervical Fusion
MeSH Terms: conditions — Facial Pain; Neck Pain; Back Pain; Klippel-Feil Syndrome | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lidocaine skin wheal (Sham Comparator): They will receive an injection of lidocaine in the skin over the area of the trigger points. While this causes a small area of numbness, it is not a trigger point injection.
  Interventions: Drug: Lidocaine skin wheal
- Trigger point injection with normal saline (Active Comparator): Trigger point injections in the rhomboid and trapezius regions with up to 20cc of 0.9% Normal Saline + intra- and postoperative standardized analgesia regimen
  Interventions: Drug: Trigger point injection with normal saline
- Trigger point injection with bupivacaine (Experimental): Trigger point injections in the rhomboid and trapezius regions with up to 20cc of 0.25% bupivacaine hydrochloride + intra- and postoperative standardized analgesia regimen
  Interventions: Drug: Trigger point injection with bupivacaine

INTERVENTIONS:
Drug: Trigger point injection with bupivacaine — Trigger point injections will be performed within an hour of arrival in post anesthesia care unit, given that the patient has adequately woken up from general anesthesia. Injections will be performed by an anesthesiology provider using a standardized technique under strict aseptic conditions. The trigger point will be located between two fingers, and a 1-2cm sterile needle with a thickness of 25 or 26 gauge inserted at 30 degrees with respect to the skin. Negative aspiration will be confirmed before injecting the study solution. The needle will be withdrawn to the subcutaneous tissue and redirected superiorly, inferiorly, laterally and medially, injecting study solution at each location. Pressure will be applied to the area to ensure hemostasis, and the area dressed with gauze and tape as needed.
  Arms: Trigger point injection with bupivacaine
Drug: Trigger point injection with normal saline — Trigger point injections will be performed within an hour of arrival in post anesthesia care unit, given that the patient has adequately woken up from general anesthesia. Injections will be performed by an anesthesiology provider using a standardized technique under strict aseptic conditions. The trigger point will be located between two fingers, and a 1-2cm sterile needle with a thickness of 25 or 26 gauge inserted at 30 degrees with respect to the skin. Negative aspiration will be confirmed before injecting the study solution. The needle will be withdrawn to the subcutaneous tissue and redirected superiorly, inferiorly, laterally and medially, injecting study solution at each location. Pressure will be applied to the area to ensure hemostasis, and the area dressed with gauze and tape as needed.
  Arms: Trigger point injection with normal saline
Drug: Lidocaine skin wheal — Patients in the control group will receive a small skin wheal of lidocaine. This will keep the patient blinded to the study group they are in since all patients will receive an injection.
  However, this skin wheal is not considered a trigger point injection.
  Arms: Lidocaine skin wheal

SUMMARY:
To achieve appropriate exposure for an anterior neck surgery (for example an Anterior Cervical Discectomy and Fusion or ACDF), patients are positioned supine with their neck extended. Due to being in this position, patients frequently complain of posterior neck stiffness and pain postoperatively in addition to the anterior incisional pain. This posterior cervical pain can be classified as myofascial pain.

Cervical myofascial pain is thought to be the result of overuse or trauma to the supporting muscles of the neck and shoulders. Trigger point injections are one of the methods used to treat myofascial pain. The trigger point injection procedure is where a physician (typically an anesthesiologist) performs an exam of the patient neck and upper back and finds areas of point tenderness. The physician will then inject a small amount of numbing medication (such as bupivacaine) into the muscle or tissue in that area.

Trigger point injections have been shown to be superior to botox injections or dry needling, and equivalent to physical therapy. However, these studies were performed on patients with chronic neck pain. There are no studies evaluating the effectiveness of trigger point injections on post anterior cervical surgery patients.

At our institution, trigger point injections with local anesthetic are used as part of a multimodal pain control regimen for post-anterior cervical surgery patients. Our hypothesis is if the addition of trigger point injections to standard of care multi-modal post-operative pain control will decrease patients' myofascial pain, and thereby decrease the amount of narcotic pain medication used.

ELIGIBILITY:
Inclusion Criteria:

* Elective anterior cervical surgery

Exclusion Criteria:

* Emergency surgery
* Local anesthetic allergy
* Long term opioid usage (not including tramadol and codeine)
* Intra-operative complication (e.g. unstable cervical spine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption in the first 6 hour period after intervention (trigger point injection/sham) | 6 hours after intervention
  Cumulative dose of opioid medications utilized in the time period. Measured in oral morphine equivalents.
Opioid consumption in the first 12 hour period after intervention (trigger point injection/sham) | 12 hours after intervention
  Cumulative dose of opioid medications utilized in the time period. Measured in oral morphine equivalents.
Opioid consumption in the first 24 hour period after intervention (trigger point injection/sham) | 24 hours after intervention
  Cumulative dose of opioid medications utilized in the time period. Measured in oral morphine equivalents.

SECONDARY OUTCOMES:
Pain score at 6 hours after intervention (trigger point injection/sham) | 6 hours after intervention
  Pain score will be assessed using visual analog scale. 0 indicates no pain and 10 indicates the worst possible pain.
Pain score at 12 hours after intervention (trigger point injection/sham) | 12 hours after intervention
  Pain score will be assessed using visual analog scale. 0 indicates no pain and 10 indicates the worst possible pain.
Pain score at 24 hours after intervention (trigger point injection/sham) | 24 hours after intervention
  Pain score will be assessed using visual analog scale. 0 indicates no pain and 10 indicates the worst possible pain.
Post-operative length of stay | Through hospital discharge, an average of 2 days
  Measured in days and hours

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No